CLINICAL TRIAL: NCT01478828
Title: Pharmacodynamic Trial of Pre-Prostatectomy Lovastatin on MYC (V-myc Myelocytomatosis Viral Oncogene Homolog) Down-Regulation in Localized Prostate Cancer
Brief Title: Pre-Prostatectomy Lovastatin on Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to an unanticipated serious adverse event.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Patrick C Walsh Prostate Cancer Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1153; NA_00048234 (Other: JHM IRB)
Record Dates: First submitted 2011-11-03; First posted 2011-11-23 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lovastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lovastatin (Experimental): After informed consent and central pathology review of the core prostate biopsy, eligible patients who decide to undergo prostatectomy at Johns Hopkins will be scheduled to receive po lovastatin following a four times a day schedule, at the starting dose of 20 mg/kg/day. Following an initial period of monitoring for safety at this entry dose level of one month, we will then accrue patients to dose de-escalation (to 1, and 10 mg/kg/day) cohorts.
  Interventions: Drug: Lovastatin

INTERVENTIONS:
Drug: Lovastatin — oral qd varying dose escalations/de-escalations
  Other Names: Altoprev®; Mevacor®

SUMMARY:
To determine the dose of continuous daily oral lovastatin needed to achieve MYC [v-myc myelocytomatosis viral oncogene homolog (avian)] down-regulation in prostatectomy specimens in intermediate-/high-risk localized prostate cancer patients.

DETAILED DESCRIPTION:
Pharmacodynamic Phase 0 trial of pre-prostatectomy lovastatin to downregulate MYC in localized prostate cancer.

Rationale: Based on available clinical and preclinical data, the investigators theorize that high-dose lovastatin therapy will decrease MYC levels in human prostate cancers shown to have MYC overexpression on biopsy.

Experimental Methods: The investigators propose a prospective, dose-finding pharmacodynamic study of lovastatin in intermediate/high-grade localized prostate cancer. The study will involve 30 eligible patients with localized prostate cancer with a Gleason sum of 7 to 10 who elect to undergo prostatectomy at Johns Hopkins. Five eligible men will be scheduled to receive oral lovastatin following a four times a day schedule, at the starting dose of 12 mg/kg/day. Patients will receive 2 weeks (14 days) of daily oral lovastatin prior to surgery. Following an initial safety monitoring period of a month, the investigators enroll at the next dose level (20 mg/kg/day). Similar dose de-escalation will continue over three more dose levels (1, 4 and 8 mg/kg/day) until 25 patients total are enrolled. Following surgery, prostatectomy specimens will undergo MYC immunohistochemistry (IHC) and compared to MYC IHC from matched biopsy samples. Pharmacodynamic efficacy (PE) will be defined as greater than 60% inhibition of MYC expression by IHC in greater than 60% of patients in prostatectomy tumor specimens compared to the matched biopsy.

Expected Results: The investigators expect lovastatin will enforce the downregulation of MYC levels in prostatectomy samples as compared to pre-lovastatin treatment core biopsy samples. The investigators also expect little toxicity to patients as reported in prior phase I and II trials using similar doses of lovastatin.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the prostate, without evidence of spread beyond to lymph nodes, bone, or visceral organs, stage T1c or higher.
2. Tumor Gleason sum of 7 (4+3 and 3+4 allowed) in at least one core, after central review of prostate biopsy at Johns Hopkins. However, in accordance with standard clinical practices, adenocarcinoma must be present in at least two discrete biopsy sections ( may vary in Gleason score).
3. Age ≥18 years of age.
4. Radical prostatectomy scheduled at Johns Hopkins.
5. Willingness to sign and ability to understand informed consent.
6. No history of treatment with any statin-class medication within 6 months of entry into the trial.
7. ECOG (Eastern Cooperative Oncology Group) performance status 0-1.
8. Adequate bone marrow, hepatic, and renal function as determined by:

WBC (white blood cells) >3,500 cells/mm3 ANC (absolute neutrophil count) >1,500 cells/mm3 Hemoglobin >9 g/dl Platelet count >100,000 cells/mm3 Serum creatinine < 2.6 mg/dl Serum bilirubin <2 mg/dl ALT (alanine aminotransferase), AST (aspartate aminotransferase), and Alkaline Phosphatase <2 times the upper limit of normal Triglycerides and total cholesterol <3 times the upper limit of normal

Exclusion Criteria:

1. Patients with evidence of metastatic prostate cancer, including bone, visceral, brain, and lymph node metastases.
2. Other histologic prostate cancers, including ductal, sarcomatous, lymphoma, small cell, and neuroendocrine tumors.
3. Uncontrolled medical conditions that could potentially increase the risk of toxicities or complications of this therapy including active liver disease, unexplained persistent elevation of serum transaminases, or medications that interfere with the metabolism of lovastatin, or gastrointestinal disease that would limit the ability to swallow or take oral medications or absorb them.
4. Concurrent malignancy other than prostate cancer.
5. Inability to provide informed consent.
6. Concomitant use of azole antifungals, cyclosporine, clarithromycin, erythromycin, fibric acid derivatives, lopinavir/ritonavir, niacin, ritonavir/saquinavir
7. Prior chemotherapy, radiation therapy, biologic therapy, or immunotherapy for prostate cancer.
8. Poor performance status (ECOG >1).
9. Prostatectomy at other hospital other than Johns Hopkins.
10. Prior history of allergy or severe reaction to statins or statin derivatives.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-07-13 (Actual); Primary Completion 2013-04-08 (Actual); Study Completion 2013-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phouc Tran, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lovastatin
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lovastatin
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Can Achieve 60% MYC Modulation Response
Description: Number of participants who achieve V-myc Myelocytomatosis Viral Oncogene Homolog (MYC) down-regulation in prostatectomy specimens in intermediate-/high-risk localized prostate cancer patients.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Lovastatin
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Number of Participants Who Experience Specific Adverse Events at Different Dosing Points Prior to Surgery.
Description: Toxicity of the different doses of continuous daily oral lovastatin in generally healthy men with prostate cancer prior to surgery.
Time Frame: 1 year
Population: Data was not collected for this outcome measure due to early study termination.
Arm/Group | Lovastatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Men With MYC Target Inhibition in Prostate Tumor Tissue
Description: Proportion of men with MYC target inhibition in prostate tumor tissue using paired tumor biopsies before and after lovastatin administration.
Time Frame: 1 year
Population: Data was not collected for this outcome measure due to early study termination.
Arm/Group | Lovastatin
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Cholesterol Level After Lovastatin Treatments.
Description: Change in cholesterol level with each tested dose of oral lovastatin.
Time Frame: 1 year
Population: Data was not collected for this outcome measure due to early study termination.
Arm/Group | Lovastatin
Number analyzed (Participants) | 0

5. Secondary Outcome: Pharmacodynamic Changes in Participants After the Pre-treatment Biopsy as Measured by Number of Participants With Target Inhibition of MYC
Description: Number of participants with target inhibition of MYC in relationship with pretreatment prostate biopsy Gleason sum, Ki-67, and degree of MYC overexpression.
Time Frame: 1 year
Population: Data was not collected for this outcome measure due to early study termination.
Arm/Group | Lovastatin
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Target Inhibition of MYC and Increased Apoptosis and Proliferation
Description: Number of participants with target inhibition of MYC and markers of increased apoptosis (cleaved caspase-3) and proliferation (Ki-67).
Time Frame: 1 year
Population: Data was not collected for this outcome measure due to early study termination.
Arm/Group | Lovastatin
Number analyzed (Participants) | 0

7. Secondary Outcome: Study Compliance as Assessed by Number of Participants Who Follow All of the Study Rules.
Time Frame: 1 year
Population: Data was not collected for this outcome measure due to early study termination.
Arm/Group | Lovastatin
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With MYC Downregulation
Description: Number of participants with MYC downregulation after high-dose lovastatin.
Time Frame: 1 year
Population: Data was not collected for this outcome measure due to early study termination.
Arm/Group | Lovastatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | Lovastatin
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovastatin (N=2)
rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) — patient was diagnosed with profound rhabdomyolysis with CK values in excess of 100,000 IU/L.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes